CLINICAL TRIAL: NCT03176849
Title: A Randomized Phase IV Control Trial of Single High Dose Oral Vitamin D3 (Stoss Therapy) in Pediatric Patients Undergoing HSCT to Prevent Vitamin D Deficiency and Insufficiency During Transplant
Brief Title: A Randomized Phase IV Control Trial of Single High Dose Oral Vitamin D3 in Pediatric Patients Undergoing HSCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Jessie Bodea, MD, Resident Physician, Phoenix Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-076
Record Dates: First submitted 2017-05-26; First posted 2017-06-06 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Vitamin D Deficiency; Stem Cell Transplant Complications; Pediatric Cancer; Blood Disorder; Pediatric Acute Myeloid Leukemia; Pediatric Acute Lymphoid Leukemia; Myelodysplastic Syndromes; Sickle Cell Anemia in Children; Aplastic Anemia; Thalassemia in Children
MeSH Terms: conditions — Vitamin D Deficiency; Neoplasms; Hematologic Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Anemia, Aplastic | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study will be randomized to either a control or intervention arm prior to the start of transplant using block randomization of blocks of 6. Those randomized to the intervention arm will receive the intervention (Stoss Therapy dosing of vitamin D) at the start of transplant followed by maintenance supplementation of vitamin D according to standard of care. Those randomized into the control arm will receive only maintenance supplementation of vitamin D according to standard of care throughout transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single, high dose oral vitamin D3 (Experimental): Patients will take a single oral dose of vitamin D3 based on age and initial vitamin D level. A patient will be classified as sufficient, insufficient, or deficient at the start of therapy. Following this dose, patients will also be given standard vitamin D3 supplementation according to current Endocrine Society Guidelines.
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Standard Vitamin D3 Supplementation
- Standard Vitamin D Supplementation (Active Comparator): Patients will be given standard vitamin D3 supplementation during transplant in accordance with standard of care per Endocrine Society Guidelines. This supplementation is based on a patient's initial vitamin D level.
  Interventions: Dietary Supplement: Standard Vitamin D3 Supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — The single, oral dose of vitamin D3 is based on patient's age and baseline 25-hydroxy-vitamin D level. Dosing is as follows: (1) For children under 3 years of age. 200000IU for those deficient, 150000IU for those insufficient, and 100000IU for those sufficient; (2) For children 3-12 years of age, 400000IU for those deficient, 350000IU for those insufficient, and 200000IU for those sufficient; (3) For children greater than 12 years of age, 600000IU for those deficient, 500000IU for those insufficient, and 300000IU for those sufficient. This is a single, one time oral dose given prior to the start of transplant.
  Arms: Single, high dose oral vitamin D3
Dietary Supplement: Standard Vitamin D3 Supplementation — Those who have sufficient vitamin D will be supplemented with 400-600IU/day of Vitamin D3 orally.
  Those who have insufficient or are deficient in vitamin D will be supplemented with 50,000IU/week of Vitamin D3 orally.

SUMMARY:
Research has suggested that children with sufficient vitamin D levels undergoing hematopoietic stem cell transplant (HSCT) have improved outcomes, including lower incidences of infection and graft-versus-host disease (GVHD), as well as overall improved survival. However, supplementation in children undergoing HSCT has shown to be a challenge using standard or aggressive supplementation strategies. The primary objective of this study is to determine the safety and efficacy of a single, high dose oral vitamin D (Stoss Therapy) at the start of transplant followed by maintenance supplementation in children undergoing HSCT.

DETAILED DESCRIPTION:
Comorbidities and complications including infection, organ system toxicity, graft-versus-host disease (GVHD) and disease recurrence are some of the biggest contributors to quality of life and mortality in children undergoing hematopoietic stem cell transplant (HSCT). Research has suggested that patients with sufficient vitamin D levels during transplant have improved outcomes, including lower incidences of infection and acute GVHD, as well as overall improved survival. Prior research has shown that chronically ill children are at risk for vitamin D deficiency, including those undergoing HSCT. Data has shown populations with as many as 70% of HSCT patients have insufficient levels of vitamin D at time of transplant. While several studies have attempted methods of vitamin D supplementation in this subset of patients, there has not been success with either standard or aggressive supplementation strategies.

Single high-dose oral vitamin D therapy, known as stoss therapy, has been used in other chronically ill children where adequate levels of vitamin D are difficult to attain. Stoss therapy suggests a single high-dose followed by maintenance dosing would be adequate to replete and maintain vitamin D levels in chronically ill children. While it has been shown to be effective with no evidence of toxicity in patients with rickets and cystic fibrosis, its safety and efficacy has not been studied in the transplant setting. However, there is an urgent need to identify a modifiable factor may reduce the occurrence and/or severity of HSCT associated complications. The overall objective of this study is to determine the effectiveness of a single, high dose oral vitamin D (Stoss Therapy) followed by maintenance supplementation in children undergoing HSCT. This change will result in a new and innovative approach to maintaining adequate vitamin D levels during pediatric HSCT, with the long term goal of reducing morbidity and mortality.

Our primary goal is to assess the safety and efficacy of a single, high dose of vitamin D followed by maintenance supplementation in children undergoing HSCT. Our secondary goal is to identify the effects of adequate vitamin D levels on early clinical outcomes such as cytokine levels, graft versus host disease, immune recovery, rejection, relapse, infection rates in pediatric HSCT patients.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients, ages 1 to 25 years of age, undergoing hematopoietic stem cell transplant at Phoenix Children's hospital
* Patients must sign an informed consent

Exclusion Criteria:

* Prior rejection of hematopoietic stem cell transplant

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Safety of Stoss Therapy | 100 days
  In order to monitor the safety of stoss therapy, patients will be monitored for any clinical signs or symptoms of hypervitaminosis D, including abdominal pain, dehydration, and fatigue. Patients will be monitored for hypercalcemia and hyperphosphatemia with weekly complete metabolic panels and serum phosphorus during the first 100 days of transplant. Patients will have repeat measurements of serum 25(OH)D levels will be obtained at Day +30 to ensure they do not have hypervitaminosis D at that time.
Efficacy of vitamin D repletion | 100 days
  All patients will have baseline serum 25(OH)D levels obtained prior to transplant. At baseline, patient will be classified as being sufficient (>30ng/mL), insufficient (21- 29ng/mL), or deficient (<20ng/mL) in serum vitamin D. All patients will then undergo treatment based on their trial arm and baseline levels of vitamin D. Patients will have repeat measurements of serum 25(OH)D levels will be obtained at Day +100 of transplant. At this time they will again be classified as being sufficient (>30ng/mL), insufficient (21- 29ng/mL), or deficient (<20ng/mL) in serum vitamin D following therapy to assess if the therapy was efficacious in repleting and maintaining their serum vitamin D level.

SECONDARY OUTCOMES:
Graft-versus-host disease | 100 days
  All incidences of GVHD will be recorded in the medical record throughout transplant as per standard of care for data extraction after Day +100
Immune Recovery | 100 days
  Immune recovery will be obtained at Day +100 as per standard of care and recorded in the medical record
Rejection | 100 days
  All incidences of rejection will be recorded in the medical record throughout transplant as per standard of care for data extraction after Day +100
Relapse | 100 days
  All incidences of relapse will be recorded in the medical record throughout transplant as per standard of care for data extraction after Day +100
Infection Rates | 100 days
  All incidences of infection will be recorded in the medical record throughout transplant as per standard of care for data extraction after Day +100
Mortality | 100 days
  All incidences of mortality will be recorded in the medical record throughout transplant as per standard of care for data extraction after Day +100

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ngwube, MD, Principal Investigator — Phoenix Children's Hospital; Kayla Burgett, Study Chair — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duncan CN, Vrooman L, Apfelbaum EM, Whitley K, Bechard L, Lehmann LE. 25-hydroxy vitamin D deficiency following pediatric hematopoietic stem cell transplant. Biol Blood Marrow Transplant. 2011 May;17(5):749-53. doi: 10.1016/j.bbmt.2010.10.009. Epub 2010 Oct 15. PMID 20951818
- [Background] Gordon CM, DePeter KC, Feldman HA, Grace E, Emans SJ. Prevalence of vitamin D deficiency among healthy adolescents. Arch Pediatr Adolesc Med. 2004 Jun;158(6):531-7. doi: 10.1001/archpedi.158.6.531. PMID 15184215
- [Background] Hansson ME, Norlin AC, Omazic B, Wikstrom AC, Bergman P, Winiarski J, Remberger M, Sundin M. Vitamin d levels affect outcome in pediatric hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2014 Oct;20(10):1537-43. doi: 10.1016/j.bbmt.2014.05.030. Epub 2014 Jun 5. PMID 24910378
- [Background] Heaney RP, Armas LA, Shary JR, Bell NH, Binkley N, Hollis BW. 25-Hydroxylation of vitamin D3: relation to circulating vitamin D3 under various input conditions. Am J Clin Nutr. 2008 Jun;87(6):1738-42. doi: 10.1093/ajcn/87.6.1738. PMID 18541563
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Misra M, Pacaud D, Petryk A, Collett-Solberg PF, Kappy M; Drug and Therapeutics Committee of the Lawson Wilkins Pediatric Endocrine Society. Vitamin D deficiency in children and its management: review of current knowledge and recommendations. Pediatrics. 2008 Aug;122(2):398-417. doi: 10.1542/peds.2007-1894. PMID 18676559
- [Background] Rosenblatt J, Bissonnette A, Ahmad R, Wu Z, Vasir B, Stevenson K, Zarwan C, Keefe W, Glotzbecker B, Mills H, Joyce R, Levine JD, Tzachanis D, Boussiotis V, Kufe D, Avigan D. Immunomodulatory effects of vitamin D: implications for GVHD. Bone Marrow Transplant. 2010 Sep;45(9):1463-8. doi: 10.1038/bmt.2009.366. Epub 2010 Jan 18. PMID 20081878
- [Background] Schlereth F, Badenhoop K. [Vitamin D : More than just a bone hormone]. Internist (Berl). 2016 Jul;57(7):646-55. doi: 10.1007/s00108-016-0082-2. German. PMID 27307163
- [Background] Shepherd D, Belessis Y, Katz T, Morton J, Field P, Jaffe A. Single high-dose oral vitamin D3 (stoss) therapy--a solution to vitamin D deficiency in children with cystic fibrosis? J Cyst Fibros. 2013 Mar;12(2):177-82. doi: 10.1016/j.jcf.2012.08.007. Epub 2012 Sep 19. PMID 22998937
- [Background] Sullivan SS, Rosen CJ, Halteman WA, Chen TC, Holick MF. Adolescent girls in Maine are at risk for vitamin D insufficiency. J Am Diet Assoc. 2005 Jun;105(6):971-4. doi: 10.1016/j.jada.2005.03.002. PMID 15942551
- [Background] Wallace G, Jodele S, Myers KC, Dandoy CE, El-Bietar J, Nelson A, Taggart CB, Daniels P, Lane A, Howell J, Teusink-Cross A, Davies SM. Vitamin D Deficiency in Pediatric Hematopoietic Stem Cell Transplantation Patients Despite Both Standard and Aggressive Supplementation. Biol Blood Marrow Transplant. 2016 Jul;22(7):1271-1274. doi: 10.1016/j.bbmt.2016.03.026. Epub 2016 Apr 1. PMID 27044905
- [Background] Wallace G, Jodele S, Howell J, Myers KC, Teusink A, Zhao X, Setchell K, Holtzapfel C, Lane A, Taggart C, Laskin BL, Davies SM. Vitamin D Deficiency and Survival in Children after Hematopoietic Stem Cell Transplant. Biol Blood Marrow Transplant. 2015 Sep;21(9):1627-31. doi: 10.1016/j.bbmt.2015.06.009. Epub 2015 Jun 18. PMID 26093045
- [Derived] Olsen B, Bodea J, Garcia A, Beebe K, Campbell C, Schwalbach C, Salzberg D, Miller H, Adams R, Mirea L, Castillo P, Horn B, Bansal S, Mohanakumar T, Ngwube A. Vitamin D Supplementation: Association With Serum Cytokines in Pediatric Hematopoietic Stem Cell Transplantation. Front Pediatr. 2022 Jul 13;10:913586. doi: 10.3389/fped.2022.913586. eCollection 2022. PMID 35911824
- [Derived] Bodea J, Beebe K, Campbell C, Salzberg D, Miller H, Adams R, Mirea L, Castillo P, Horn B, Bansal S, Mohanakumar T, Ngwube A. Stoss therapy is safe for treatment of vitamin D deficiency in pediatric patients undergoing HSCT. Bone Marrow Transplant. 2021 Sep;56(9):2137-2143. doi: 10.1038/s41409-021-01294-x. Epub 2021 Apr 19. PMID 33875811
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- See also: More information about clinical trials at Phoenix Children's Hospital's Center for Cancer and Blood Disorders — https://www.phoenixchildrens.org/research-institute/clinical-research/clinical-trial-listing